CLINICAL TRIAL: NCT04136912
Title: High Frame Rate 3-D Super Resolution Ultrasound Microvascular Imaging
Brief Title: 3-D Super Resolution Ultrasound Microvascular Imaging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Grant ended
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC1915; R01CA220681 (NIH)
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Thyroid Cancer
Keywords: Cancer Screening
MeSH Terms: conditions — Breast Neoplasms; Thyroid Neoplasms | interventions — perflutren

STUDY DESIGN:
Intervention Model Description: Acoustic angiography is a new type of contrast enhanced ultrasound imaging which is specifically sensitive to microvascular structure and density.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Breast Imaging Cohort (Experimental): A total of 15 women with known breast lesions that are already scheduled to undergo a clinical biopsy
  Interventions: Drug: Definity; Device: Acoustic Angiography
- Thyroid Imaging Cohort (Experimental): A total of 15 participants with known thyroid lesions that are already scheduled to undergo a clinical biopsy
  Interventions: Drug: Definity; Device: Acoustic Angiography
- Healthy Volunteers Cohort (Experimental): A total of 15 participants will be included to optimize imaging parameters.
  Interventions: Drug: Definity; Device: Acoustic Angiography

INTERVENTIONS:
Drug: Definity — Perflutren will be administered in split doses using the dosing range and administration type IV bolus) within the perflutren prescribing information. When administered as a bolus, the package insert recommends 10 uL/kg patient weight administered within 30-60 seconds, followed by a 10mL saline flush with a second dose of 10 uL/kg patient weight 30 minutes following the first dose, if needed.
  Other Names: perflutren
Device: Acoustic Angiography — Acoustic angiography imaging involves a research ultrasound scanner as well as conventional b-mode ultrasound to guide the location of the imaging. The conventional ultrasound will be conducted just prior to the acoustic angiography for localization. Imaging will be performed within the package insert guidelines for ultrasound system mechanical index (a measurement of output power) when imaging perflutren contrast agent (less than 0.8).
  Acoustic angiography imaging will be performed by trained medical personnel using mild compression to eliminate motion. Total imaging time is estimated to be less than 15 minutes.

SUMMARY:
This is a 3-arm single center study of 45 patients. These cohorts will include 15 breast patients scheduled to undergo a biopsy, and 15 thyroid patients scheduled to undergo fine needle aspiration, biopsy, or thyroidectomy that consent to undergo an acoustic angiography in conjunction with b-mode ultrasound prior to their scheduled biopsy. Prior to imaging clinical patients, the third arm will include 15 healthy volunteers that will be imaged to optimize imaging parameters.

DETAILED DESCRIPTION:
Increasing the sensitivity and specificity of diagnostic imaging in patients at high risk for breast or thyroid cancer could provide substantial clinical benefit by improving diagnosis, preventing over-treatment, and reducing healthcare costs. Acoustic angiography is a new type of contrast enhanced ultrasound imaging which is specifically sensitive to microvascular structure and density. It evaluates tumor micro-vasculature and may provide a powerful prognostic tool for the diagnosis of breast cancer, and eventually for treatment evaluation.

ELIGIBILITY:
Healthy Volunteers

Inclusion Criteria

* Able to provide informed consent
* Negative urine pregnancy test in women of child-bearing potential

Exclusion Criteria

* Institutionalized subject (prisoner or nursing home patient)
* Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD)
* Known hypersensitivity to perflutren lipid (Definity®)
* Active cardiac disease including any of the following:

  * Severe congestive heart failure
  * Unstable angina.
  * Severe arrhythmia
  * Myocardial infarction within 14 days prior to the date of proposed Definity® administration.
  * Pulmonary hypertension
  * Cardiac shunts

Breast Imaging Patients

Inclusion Criteria

* Women
* Patient had a diagnostic breast ultrasound study performed at UNC
* Scheduled for a core needle or surgical breast biopsy of at least one breast lesion that is 2 cm or less in size and 3 cm in depth from the skin surface
* Able to provide informed consent
* Negative urine pregnancy test in women of child-bearing potential
* BIRADS score of 4 or 5.

Exclusion Criteria

* Male
* Institutionalized subject (prisoner or nursing home patient)
* Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD)
* Sonographically visible breast lesion larger than 2cm or greater than 3cm in depth from the skin surface
* Known hypersensitivity to perflutren lipid (Definity®)
* Active cardiac disease including any of the following:

  * Severe congestive heart failure
  * Unstable angina.
  * Severe arrhythmia
  * Myocardial infarction within 14 days prior to the date of proposed Definity® administration.
  * Pulmonary hypertension
  * Cardiac shunts

Thyroid Imaging Patients Inclusion Criteria

* Patient had a diagnostic thyroid ultrasound study performed at UNC
* TIRADS risk score of 4c or 5
* Scheduled for a core needle or surgical thyroid biopsy, fine needle aspiration, or thyroidectomy of at least one sonographically visible thyroid lesion that is 3 cm in depth from the skin surface
* Able to provide informed consent
* Negative urine pregnancy test in women of child-bearing potential

Exclusion Criteria

* Institutionalized subject (prisoner or nursing home patient)
* Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD)
* Known hypersensitivity to perflutren lipid (Definity®)
* Active cardiac disease including any of the following:

  * Severe congestive heart failure
  * Unstable angina.
  * Severe arrhythmia
  * Myocardial infarction within 14 days prior to the date of proposed Definity® administration.
  * Pulmonary hypertension
  * Cardiac shunts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Lee, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Univeristy of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results
Supporting Information: Study Protocol
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: An investigator who proposes to use the data must have approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a North Carolina cancer center from 04/11/2022 to 08/01/2024, with enrollment occurring between 05/26/2022 and 08/01/2024. The study closed before reaching its target enrollment due to insufficient funding.
Pre-assignment Details: Twenty-eight participants consented to the study; one was ineligible and not enrolled. No participants were enrolled in Arm 2 (Thyroid Imaging). Twelve were enrolled in Arm 1 (Breast Imaging), and fifteen in Arm 3 (Healthy Volunteers).
Groups:
- Breast Imaging Cohort: Women with known breast lesions that are already scheduled to undergo a clinical biopsy.
- Thyroid Imaging Cohort: Participants with known thyroid lesions that are already scheduled to undergo a clinical biopsy.
Period: Overall Study
Arm/Group | Breast Imaging Cohort | Thyroid Imaging Cohort | Healthy Volunteers Cohort
Started | 12 | 0 | 15
Completed | 12 | 0 | 13
Not Completed | 0 | 0 | 2
Not completed — Operational reasons | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All eligible participants who consented were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Imaging Cohort | Thyroid Imaging Cohort | Healthy Volunteers Cohort | Total
Number analyzed (Participants) | 12 | 0 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.83 (18.35) |  | 29.73 (12.57) | 41.17 (18.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 0 | 15 | 27
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 0 | 15 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 8 | 0 | 14 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 |  | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Acoustic Angiography; Breast Imaging
Description: The sensitivity of Acoustic Angiography in the analysis of known breast lesions will be evaluated by comparing image analyses to the pathological results for these lesions.
  Sensitivity (%) = True Positives (TP)+False Negatives (FN)True Positives (TP)
Time Frame: Baseline
Population: Patients with known breast lesion.
Measure: Number; unit: percentage
Arm/Group | Breast Imaging Cohort
Number analyzed (Participants) | 12
percentage | 50

2. Primary Outcome: Specificity of Acoustic Angiography; Breast Imaging (Percent of Negative Scans)
Description: Specificity of Acoustic Angiography in the analysis of known breast lesions will be evaluated by comparing image analyses to the pathological results for these lesions. Specificity was calculated based on the formula, which is true negative / (true negative + false positive).
Time Frame: Baseline
Population: Patient with known breast lesion.
Measure: Number; unit: percentage of benign lesion
Arm/Group | Breast Imaging Cohort
Number analyzed (Participants) | 12
percentage of benign lesion | 67

3. Primary Outcome: Sensitivity of Acoustic Angiography; Thyroid Imaging (Percent of Positive Scans)
Description: Sensitivity of Acoustic Angiography in the analysis of know thyroid lesions will be evaluated by comparing image analyses to the pathological results for these lesions. The study closed early due to insufficient funding and did not reach target enrollment. No participants were enrolled in Arm 2 (Thyroid Imaging); therefore, no outcome measure results are available.
Time Frame: Baseline
Arm/Group | Thyroid Imaging Cohort
Number analyzed (Participants) | 0

4. Primary Outcome: Specificity of Acoustic Angiography; Thyroid Imaging (Percent of Negative Scans)
Description: Specificity of Acoustic Angiography in the analysis of known thyroid lesions will be evaluated by comparing image analyses to the pathological results for these lesions. The study closed early due to insufficient funding and did not reach target enrollment. No participants were enrolled in Arm 2 (Thyroid Imaging); therefore, no outcome measure results are available.
Time Frame: Baseline
Arm/Group | Thyroid Imaging Cohort
Number analyzed (Participants) | 0

5. Secondary Outcome: Area Under the Curve of Acoustic Angiography (Arbitrary Units)
Description: To compare the area under the curve (AUC) of acoustic angiography to the AUC of the B-mode ultrasound. Readers assigned a malignancy likelihood score from 1 to 5, with 1 likely benign to 5 likely malignant. An AUC was then calculated based on these scores. The Receiver operating curve (ROC ) was then plotted from this curve, and the AUC was estimated from the ROC curve.
Time Frame: Baseline
Population: Patient with a known breast lesion.
Measure: Number; unit: percentage of probability
Arm/Group | Breast Imaging Cohort
Number analyzed (Participants) | 12
percentage of probability | 50

6. Secondary Outcome: Radiologist Preference (Arbitrary Units)
Description: To compare radiologist preference of acoustic angiography (AA) to conventional b-mode ultrasound, for each lesion characteristics which are shape, margins, and vascularity, were examined. Radiologists rated their preferences on a Likert scale from 1 to 5, with 1 strongly preferring conventional ultrasound and 5 strongly preferring AA.
  Shape, margin, and vascularity values appear to represent mean or median rather than counts. We should select either the mean or the median and provide the standard deviation, which will be 0 if all radiologists assign the same score.
Time Frame: Baseline
Population: Patients with a known breast lesion.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Breast Imaging Cohort
Number analyzed (Participants) | 12
score on a scale
  shape | 1 (0)
  margin | 1 (0)
  vascularity | 5 (0)

7. Secondary Outcome: Sensitivity of Acoustic Angiography Compared to Conventional Ultrasound: Breast (Arbitrary Units)
Description: Sensitivity of Acoustic Angiography relative to conventional ultrasound in the analysis of known breast lesions will be evaluated by comparing image analyses to the pathological results for these lesions for both modalities. Sensitivity was calculated based on the formula, which is true positive / (true positive + false negative). The ratio between the sensitivity of AA over the sensitivity of conventional ultrasound was then calculated.
Time Frame: Baseline
Population: Patients with malignant breast lesion(s).
Measure: Number; unit: ratio
Arm/Group | Breast Imaging Cohort
Number analyzed (Participants) | 12
ratio | 1.2

8. Secondary Outcome: Specificity of Acoustic Angiography Compared to Conventional Ultrasound: Breast (Arbitrary Units)
Description: Specificity of Acoustic Angiography (AA) and conventional ultrasound in the analysis of known breast lesions will be evaluated by comparing image analyses to the pathological results for these lesions for each modality. Specificity was calculated based on the formula, which is true negative / (true negative + false positive). The ratio between the sensitivity of AA over the sensitivity of conventional ultrasound was then calculated.
Time Frame: Baseline
Population: Patients with known breast lesion(s).
Measure: Number; unit: ratio
Arm/Group | Breast Imaging Cohort
Number analyzed (Participants) | 12
ratio | 0.86

9. Secondary Outcome: Sensitivity of Acoustic Angiography Compared to Conventional Ultrasound: Thyroid (Arbitrary Units)
Description: To compare (using a reader study) the sensitivity of acoustic angiography to the sensitivity of conventional b-mode ultrasound in evaluation of known thyroid lesions for predicting malignancy. The study closed early due to insufficient funding and did not reach target enrollment. No participants were enrolled in Arm 2 (Thyroid Imaging); therefore, no outcome measure results are available.
Time Frame: Baseline
Arm/Group | Thyroid Imaging Cohort
Number analyzed (Participants) | 0

10. Secondary Outcome: Specificity of Acoustic Angiography Compared to Conventional Ultrasound: Thyroid (Arbitrary Units)
Description: To compare (using a reader study) the specificity of acoustic angiography to the specificity of conventional b-mode ultrasound in evaluation of known thyroid lesions for predicting malignancy. The study closed early due to insufficient funding and did not reach target enrollment. No participants were enrolled in Arm 2 (Thyroid Imaging); therefore, no outcome measure results are available.
Time Frame: Calculated once all imaging is complete [Anticipated 1.5 years]
Arm/Group | Thyroid Imaging Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the day of imaging.
Description: Adverse events were graded according to CTCAE on the day of research imaging.
Groups:
- Breast Imaging Cohort: Women with known breast lesions that are already scheduled to undergo a clinical biopsy, and acoustic angiography imaging will be performed by trained medical personnel using mild compression to eliminate motion.
- Thyroid Imaging Cohort: Participants with known thyroid lesions that are already scheduled to undergo a clinical biopsy and acoustic angiography imaging will be performed by trained medical personnel using mild compression to eliminate motion.
- Healthy Volunteers Cohort: Participants will be included to optimize imaging parameters. Acoustic angiography imaging will be performed by trained medical personnel using mild compression to eliminate motion.
Arm/Group | Breast Imaging Cohort | Thyroid Imaging Cohort | Healthy Volunteers Cohort
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/0 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/0 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/0 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Breast Imaging Cohort (N=12) | Thyroid Imaging Cohort (N=0) | Healthy Volunteers Cohort (N=15)
flushing (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT04136912/Prot_SAP_000.pdf